CLINICAL TRIAL: NCT04335227
Title: Yoga Therapy and Aerobic Exercise on Anti-Mullerian Hormone and Other Biochemical Markers in Young Women With Polycystic Ovary Syndrome
Brief Title: Yoga Therapy and Aerobic Exercise on Anti-Mullerian Hormone in Young Women With Polycystic Ovary Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Maharishi Markendeswar University (Deemed to be University) (Other)
Responsible Party: Principal Investigator, Asir John Samuel, Associate Professor, Maharishi Markendeswar University (Deemed to be University)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MMDU/IEC/141E
Record Dates: First submitted 2020-03-27; First posted 2020-04-06 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Polycystic Ovary Syndrome; Anti-Mullerian Hormone Deficiency; Female Infertility Endocrine
Keywords: Yoga therapy; Aerobic exercise training; Aerobic exercise; Aerobic training; Polycystic ovary syndrome; Antimullerian hormone
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Diet

STUDY DESIGN:
Intervention Model Description: Recruited female with PCOS with 128 female with PCOS will be randomly divided into four parallel groups, yoga therapy (YT) group, aerobic exercise (AE) group, combined YT and AE (cYTAE) group and control group
Who Masked: Outcomes Assessor
Masking Description: Lab technician who test the blood samples of the female with Polycystic Ovary Syndrome (PCOS) will be blinded to the trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Yoga therapy group (Experimental): Structured yoga therapy program for 60 minutes six days per week for 12 weeks and nutritional management uniquely prepared by dietitian
  Interventions: Other: Structured yoga therapy program
- Aerobic exercise group (Experimental): Aerobic training of moderate intensity for 30-60 minutes six days per week for 12 weeks and nutritional management uniquely prepared by dietitian
  Interventions: Other: Aerobic exercise training program
- Combined yoga therapy and aerobic exercise group (Experimental): Combined yoga therapy for three days and vigorous aerobic exercise program for three days with nutritional management uniquely prepared by dietitian
  Interventions: Other: Combined yoga and aerobic training program
- Control group (Active Comparator): Nutritional management uniquely prepared by dietitian
  Interventions: Other: Nutritional management

INTERVENTIONS:
Other: Structured yoga therapy program — Structured yoga therapy prepared according to traditional yoga scriptures of Patanjali yoga sutras will be administered to 32 females with PCOS. The structured yoga therapy which includes, Surya Namaskara (Sun Salutation) and asanas performed in four positions, standing, sitting, supine and prone for total duration of 60 minutes. In addition to this, they will be asked to undergo nutritional management uniquely prepared by dietitian
  Arms: Yoga therapy group
Other: Aerobic exercise training program — Thirty two females with PCOS in aerobic exercise (AE) group will be subjected to aerobic training of moderate intensity for 30-60 minutes six days per week for 12 weeks, in the light of guidelines framed by American College of Sports Medicine (ACSM). Aerobic exercise volume for each female recruited will be set at greater than 500 and up to 1000 MET-min/week, which will be approximately equal to 1000 kcal/week. They will be made sure that they exercise for minimum duration of 150 min/week and thereby covering 5400 to 7900 steps/day in pedometer readings. In addition to this, they will be asked to undergo nutritional management uniquely prepared by dietitian
  Arms: Aerobic exercise group
Other: Combined yoga and aerobic training program — Thirty two females with PCOS in combined yoga therapy and aerobic exercise (cYTAE) group will be subjected to three days of structured yoga therapy and three days of aerobic training of vigorous intensity. In addition to this, they will be asked to undergo nutritional management uniquely prepared by dietitian
  Arms: Combined yoga therapy and aerobic exercise group
Other: Nutritional management — Thirty two females with PCOS will be asked to undergo only nutritional management uniquely prepared by dietitian
  Arms: Control group

SUMMARY:
Weight loss and lifestyle modifications are much required in women with Polycystic ovarian syndrome (PCOS). Yoga has gained great importance as an alternate medicine in recent years which is helpful in lifestyle modifications. Weight loss can be achieved by regular aerobic activity. In recent years, excessive production of anti-mullerian hormone (AMH) has been considered as the etiology of PCOS. AMH is also emerging as a diagnostic and screening tool for PCOS. Effect of yoga therapy on adolescent girls have proved to be effective. But, researches on young women undergoing yoga therapy and combined effect of aerobic exercise and yoga therapy are still lacking. Hence, the investigators aimed t o establish the benefits of yoga therapy and aerobic exercise on Anti-Mullerian Hormone and other biochemical markers in young women with polycystic ovary syndrome.

DETAILED DESCRIPTION:
A total of 128 female with PCOS will be recruited by the simple random sampling (random number generator) to participate in randomized, single blind randomized controlled, study. Recruited patients with 128 female with PCOS will be randomly divided into four groups, yoga therapy (YT) group, aerobic exercise (AE) group, combined YT and AE (cYTAE) group and control group. Duration of the intervention will be 60 minutes in one session for 6 days/week for 12 weeks. Thus, each women with PCOS will receive 72 sessions in total, except in control group. Anti-Müllerian hormone (AMH) and other biochemical markers such as, Follicle-stimulating hormone (FSH), Luteinizing hormone (LH), Testosterone, Prolactin, Thyroid-stimulating hormone (TSH) Ultrasensitive, Dehydroepiandrosterone sulfate (DHEAS), insulin fasting, glucose fasting, HOMA-IR (Homeostatic Model Assessment for Insulin Resistance) and the lipid profiles which includes, total cholesterol, High-density lipoprotein cholesterol (HDL-C), Low-density lipoprotein cholesterol (LDL-C) and serum triglycerides. In addition to the above biochemical markers, transvaginal ultrasound to estimate antral follicle count (AFC) will be recorded at baseline and at the end of 12-week post-intervention period. Following the 12-week intervention, follow-up of another 12-week will be carried out to determine the retention of treatment effects.

ELIGIBILITY:
Inclusion Criteria:

* Female in age between 18 and 30 years
* Female with at least two-thirds of the features listed in the Rotterdam criteria for PCOS were included in the study
* Oligomenorrhea or amenorrhea (an absence of menstruation for 45 or more days and/or fewer than 9 menses per year)
* Hyperandrogenism (a score of 8 or higher ( ≥ 8) on the modified Ferriman-Gallwey scale)
* Polycystic ovaries (presence of more than 12 cysts < 9 mm in diameter in single ovary, usually combined with an ovarian volume > 10 ml

Exclusion Criteria:

* On regular hormonal treatment
* Oral contraceptives
* Insulin-sensitizing agents in the previous 6 weeks
* Smoking in less than 48 hours
* Alcohol in less than 48 hours
* History of thyroid abnormalities
* Practicing regular yoga asanas and pranayama
* Regular aerobic training program

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female with polycystic ovarian syndrome
Enrollment: 128 (Estimated)
Dates: Start 2021-11-14 (Estimated); Primary Completion 2023-03-12 (Estimated); Study Completion 2023-04-14 (Estimated)

PRIMARY OUTCOMES:
Serum Anti-Mullerian hormone Concentration | Change from Baseline Serum Anti-Mullerian hormone Concentration at 12 weeks
  Serum Anti-Mullerian hormone will be determined by blinded lab technician

SECONDARY OUTCOMES:
Antral follicle count | Change from Baseline Antral follicle count at 12 weeks
  Antral follicle count will be determined by blinded gynaecologist
Serum Follicle-stimulating hormone Concentration | Change from Baseline Serum Follicle-stimulating hormone Concentration at 12 weeks
  Serum Follicle-stimulating hormone will be determined by blinded lab technician
Serum Luteinizing hormone Concentration | Change from Baseline Serum Luteinizing hormone Concentration at 12 weeks
  Serum Luteinizing hormone will be determined by blinded lab technician
Serum Testosterone Concentration | Change from Baseline Serum Testosterone Concentration at 12 weeks
  Serum Testosterone will be determined by blinded lab technician
Serum Prolactin Concentration | Change from Baseline Serum Prolactin Concentration at 12 weeks
  Serum Prolactin will be determined by blinded lab technician
Serum Thyroid-stimulating hormone Concentration | Change from Baseline Serum Thyroid-stimulating hormone Concentration at 12 weeks
  Serum Thyroid-stimulating hormone will be determined by blinded lab technician
Serum Dehydroepiandrosterone sulfate Concentration | Change from Baseline Serum Dehydroepiandrosterone sulfate Concentration at 12 weeks
  Serum Dehydroepiandrosterone sulfate will be determined by blinded lab technician
Serum Insulin fasting Concentration | Change from Baseline Serum Insulin fasting Concentration at 12 weeks
  Serum Insulin fasting will be determined by blinded lab technician
Serum Glucose fasting Concentration | Change from Baseline Serum Glucose fasting Concentration at 12 weeks
  Serum Glucose fasting will be determined by blinded lab technician
Homeostatic Model Assessment for Insulin Resistance | Change from Baseline Homeostatic Model Assessment for Insulin Resistance at 12 weeks
  Homeostatic Model Assessment for Insulin Resistance will be determined by blinded lab technician
Concentration of Lipid profiles in serum | Change from Baseline Concentration of Lipid profiles in serum at 12 weeks
  Serum total cholesterol, Serum High-density lipoprotein cholesterol, Serum Low-density lipoprotein cholesterol and serum triglycerides

CONTACTS AND LOCATIONS:
Overall Officials: Asir J Samuel, MPT, PhD, Principal Investigator — Maharishi Markandeshwar Institute of physiotherapy and Rehabilitation, Mullana; Unmesh Santpur, MBBS, MD, Study Director — Maharishi Markandeshwar Institute of Medical Sciences and Research, Mullana; Kiranjeet Kaur, MBBS, MD, Study Chair — Maharishi Markandeshwar Medical College & Hospital, Solan
Locations (2):
- India (2):
  - Maharishi Markandeshwar Hospital, Mullana, Ambāla, Haryana
  - Maharishi Markandeshwar Medical College & Hospital, Kumarhatti, Solan, Himachal Pradesh

IPD SHARING:
Plan to Share IPD: No
Not now